CLINICAL TRIAL: NCT02181335
Title: A Twelve-week, Efficacy and Safety Study Comparing Respimat ® Budesonide (100 and 200 mcg, 2 Puffs Bid) With Turbohaler ® Budesonide (200 mcg, 2 Puffs Bid) in Symptomatic Adult Moderate to Severe Asthmatic Requiring Inhaled Corticosteroids and Bronchodilator Therapy.
Brief Title: Efficacy and Safety Study Comparing Respimat ® Budesonide With Turbohaler ® Budesonide in Symptomatic Adult Moderate to Severe Asthmatics Requiring Inhaled Corticosteroids and Bronchodilator Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1047.16
Record Dates: First submitted 2014-07-02; First posted 2014-07-03 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (3):
- Respimat ® Budesonide low dose + Turbohaler® Placebo (Experimental)
  Interventions: Drug: Respimat® Budesonide low dose; Drug: Placebo
- Respimat ® Budesonide high dose + Turbohaler® Placebo (Experimental)
  Interventions: Drug: Respimat® Budesonide high dose; Drug: Placebo
- Turbohaler® Budesonide + Respimat Placebo® (Active Comparator)
  Interventions: Drug: Turbohaler® Budesonide; Drug: Placebo

INTERVENTIONS:
Drug: Respimat® Budesonide low dose
  Arms: Respimat ® Budesonide low dose + Turbohaler® Placebo
Drug: Respimat® Budesonide high dose
  Arms: Respimat ® Budesonide high dose + Turbohaler® Placebo
Drug: Turbohaler® Budesonide
  Arms: Turbohaler® Budesonide + Respimat Placebo®
Drug: Placebo

SUMMARY:
To establish that at least one of the two doses of Budesonide, as an ethanolic solution inhaled from the Respimat ® inhaler (100 and 200 mcg, 2 puffs bid) for a 12-week study period in symptomatic moderate to severe asthmatic patients, gives a therapeutic response, which is not inferior to that obtained from the dose of Budesonide inhaled from the Turbohaler ® (200 mcg, 2 puffs bid) and that the safety profile is at least as good

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex aged 18 - 65 years (inclusive)
* Non-smokers or ex smokers. HAVING stopped smoking >= 1 year prior to screening and with a smoking history of <= 10 pack years
* Diagnosis of MODERATE to SEVERE bronchial asthma with a duration of at least 6 months with the inclusion criteria 4 plus 5 and a diagnosis of asthma according to the WHO guidelines for at least one year
* Increase of asthma symptoms (wheeze, cough, shortness of breath, chest tightness) when exposure to any of the following stimuli: cold, dry air, dust, smoke, exercise and allergens
* Patients on a stable dosage of either

  * 800 mcg <= BDP (beclomethasone dipropionate) <= 1600 mcg daily or other inhaled steroid with or without inhaled long acting β2-agonists or oral xanthines at screening visit 1 for the past 4 weeks and short acting β2-agonists prn for the past 6 weeks or
  * 400 mcg <= BDP < 800 mcg daily or other inhaled steroid and inhaled long-acting β2-agonists (or oral xanthines), at screening visit 1 for the past 4 weeks and short acting β2-agonists prn for the past 6 weeks
* FEV1 >= 60% but <= 90 % predicted normal at visit 1 after withholding respiratory drugs as per section 4.2.1. Predicted normal values are based on the guidelines for standardized function testing of the European Community for Coal and Steel (ECCS)

  * Males: FEV1 pred. (L) = 4.30 x Height (m) - 0.029 x Age (yrs) - 2.49
  * Females: FEV1 pred. (L) = 3.95 x Height (m) - 0025 x Age (yrs) - 2.60
* Patient must demonstrate an improvement in FEV 1 >= 12% above baseline and an absolute change of at least 200 ml within 30 minutes after administration of two puffs of salbutamol MDI (metered dose inhaler) (100 mcg per puff). Historical data within the previous 6 months are acceptable
* Patients must be able to be trained in the proper use of MDI, Turbohaler® and Respimat® and to perform technically satisfactory pulmonary function tests
* Patients must be willing and be able to give informed written consent prior to participation in the trial i.e. prior to pre-study wash-out of their usual pulmonary medications and are willing and able to complete the entire study as described in the protocol

Exclusion Criteria:

* Patients with a history of seasonal exacerbation of asthma suggesting seasonal asthma which would not be controlled by medication allowed in the protocol (see 4.2.2) and likely to occur during the time period that the patients will be in the study
* History of cardiovascular, renal, neurologic, liver, immunologic or endocrine dysfunction if they are clinically significant. A clinically significant disease is defined as one which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients with a recent history (<= 1 year) of myocardial infarction and/or (<= 3 years) of heart failure or patients with any cardiac arrhythmia requiring drug therapy
* History of cancer within the past 5 years excluding treated basal cell carcinoma
* Patients with current psychiatric disorders which would interfere with the conduct of the trial
* Patients with history or presence of glaucoma and/or posterior subcapsular cataracts
* Patients who have undergone thoracotomy with pulmonary resection. Patients with a history of thoracotomy for other reasons should be evaluated as per exclusion criteria
* Patients with active tuberculosis with indication for treatment
* Patients with a history of cystic fibrosis, bronchiectasis, chronic bronchitis or emphysema
* Patients with active rhinitis requiring treatment with intranasal steroids and/or ketotifen
* Patients with upper respiratory tract infection in the past 6 weeks prior to screening visit 1 resulting in exacerbation of asthma symptoms
* Patients with unstable asthma as defined by any of the following: having required hospitalization for asthma exacerbation in the past 6 months, or a history of life-threatening asthma exacerbation resulted in respiratory failure and requiring intubation or ICU admission of longer than 24 hours in the past 5 years
* Patients with clinically signification abnormal baseline haematology, blood chemistry or urinalysis (if the abnormality defines a disease listed as an exclusion criterion)
* Patients with any of the abnormal laboratory values below:

  * SGOT (serum glutamate oxaloacetate transaminase) > 200% of the upper limit of the normal range
  * SGPT (serum glutamate pyruvate transaminase) > 200% of the upper limit of the normal range
  * Creatinine > 125% of the upper limit of the normal range
  * Bilirubin > 150% of the upper limit of the normal range, with the exception of Gilbert's disease will be excluded regardless of the clinical condition
* Patients with known intolerance hypersensitivity to one of the aerosolized products including inhaled steroids (budesonide and beclomethasone dipropionate), salbutamol, ethylenediaminetetraacetic acid, ethanol, citric or oleic acid
* Patients using oral or other systemic (intramuscular or intravenous) corticosteroids in the past 8 weeks or other potent immunosuppressant (i.e. methotrexate) medication in the past 3 months
* Patients using beta blocker therapy, ACE inhibitors (an exception was provided if the ACE inhibitor have been at a stable dose for six months with no reported incidence of cough) monoamine oxidase inhibitors, tricyclic antidepressants, cromolyn or nedocromil sodium, ketotifen, astemizole or any other antihistamine drug, or a combination of an inhaled long acting β2-agonist plus oral xanthine or having received an influenza vaccine within 1 week of Screening Visit 1
* Patients on nebulised β2-agonists, anticholinergics or steroids in the 4 weeks before screening visit 1
* If a patient is on allergen desensitization therapy, this should have been as a maintenance dose for the previous 3 months and continued throughout the treatment period
* Unstable respiratory medication dosage in the last 4 weeks prior to screening visit 1
* Patients with a significant history and/or active alcohol or drug abuse. Significant is defined as that which in the opinion of the investigator may either put the patient at risk because of participation in the study or may influence the results of the study or the patient's ability to participate in the study
* Patients who have taken any investigational drug, one month or six half-lives (whichever is greater) prior to the Screening Visit
* Pregnant or nursing women and sexually active women with childbearing potential not using a medically approved method of contraception (i.e. oral contraceptives, intrauterine devices, diaphragm, Norplant® or double-barrier)
* Previous participation in the randomised period of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 1998-10; Primary Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Change in mean weekly morning pre-dose Peak Expiratory Flow Rate (a.m. PEFR) | Day1, 15, 29, 43, 57, 71, 85 (before intake of inhaled medication)

SECONDARY OUTCOMES:
Change in Forced Expiratory Volume in one second (FEV1) | Baseline, Day1, 15, 29, 43, 57, 71, 85
Change in Forced Vital Capacity (FVC) | Baseline, Day1, 15, 29, 43, 57, 71, 85
Change in Peak Expiratory Flow Rate (PEFR) | Baseline, Day1, 15, 29, 43, 57, 71, 85
Changes in Mean weekly evening pre-dose PEFR (p.m. PEFR) | Day1, 15, 29, 43, 57, 71, 85 (before intake of inhaled medication)
Daily puffs of β2-agonists usage | up to 85 days
Diurnal and nocturnal asthma symptom score | up to 85 days
Symptoms free days and/or nights | up to 85 days
Withdrawal due to moderate or severe asthma exacerbation | up to 85 days
Change in Forced expiratory flow at 25-75% of vital capacity (FEF 25-75%) | Baseline, Day1, 15, 29, 43, 57, 71, 85
Change in systolic blood pressure | Baseline, Day1, 15, 29, 43, 57, 71, 85
Change in pulse rate | Baseline, Day1, 15, 29, 43, 57, 71, 85
Change from baseline in 12-lead electrocardiogram (ECG) | Baseline, Day 85
Changes from baseline in laboratory parameters | Baseline, Day 85
Occurence of adverse events | up to 85 days
Incidence of administration related bronchoconstriction at first and last dose | Day 1, Day 85
Markers of bone formation - Plasma osteocalcin levels (sub-group of patients) | Day 1, Day 85
Markers of bone formation - Bone alkaline phosphatase (sub-group of patients) | Day 1, Day 85
Markers of bone formation - serum calcium (all study population) | Day 1, Day 85
Markers of bone formation - serum phosphate (all study population) | Day 1, Day 85
Markers of bone formation - serum procollagen I (sub-group of patients) | Day 1, Day 85
Markers of bone dissolution - Urine deoxypyridiline (subset of patients) | Day 1, Day 85
Serum cortisol levels (a.m.) - (subset of study population) | Day 1, 29, 57, 85
10 hour urinary free cortisol/creatinine ratio (subset of study population) | Day 1, 29, 57, 85
Oral Candidiasis (quantitative assessment) | up to 85 days
Incidence of hoarseness of voice | up to 85 days
Incidence of sore throat | up to 85 days
Markers of bone formation - Alkaline phosphatase (all study population) | Day1, Day 85